CLINICAL TRIAL: NCT05381467
Title: The Bone Shielding Versus Dual Zone Concept in Treating Thin Walled Fresh Extraction Sockets With Immediate Implant Placement Soft and Hard Tissue Changes A Randomized Clinical Trial
Brief Title: Evaluation of Immediate Implant Placement In The Esthetic Zone Using the Bone Shielding Concept Versus Dual Zone Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nesma Mohamed Fouad Shemais, PhD holder Lecturer in the department of Oral Medicine & Periodontology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAN.1
Record Dates: First submitted 2022-05-11; First posted 2022-05-19 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Immediate Implants; Alveolar Bone Loss; Dual Zone Technique; the Bone Shielding Concept; Esthetic Zone
Keywords: esthetic zone; soft tissue augmentation
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- immediate implant placement with The Dual-Zone Therapeutic Concept (Active Comparator)
  Interventions: Procedure: immediate implant placement with The Dual-Zone Therapeutic Concept
- Immediate implant placement with the bone shielding concept (Experimental)
  Interventions: Procedure: Immediate implant placement with the bone shielding concept

INTERVENTIONS:
Procedure: immediate implant placement with The Dual-Zone Therapeutic Concept — After tooth removal, implant placement, bone grafting, and screw retained provisional restoration, the contour of the ridge can change. Using dual zone grafting was claimed to minimize contour change associated with immediate anterior implants. In this technique. The implant should be placed in an optimal 3 dimensional mode . Xenograft, will be used in the gap to graft the bone and tissue zones, . The graft material helps serve as a scaffold to maintain hard- and soft-tissue volume as well as blood clot for initial healing.
  Arms: immediate implant placement with The Dual-Zone Therapeutic Concept
Procedure: Immediate implant placement with the bone shielding concept — After atraumatic tooth extraction using periotomes and luxators , socket curettage and cleaning simultaneously using an irrigation curette will be performed. Sulcular dissection of the attached tissue close to the socket orifice incisal and apically will be done using periotome to create a tunnel via the socket orifice. Dental implant will be placed. complete access of the labial plate of bone where all the regenerative materials will be performed to have the bone sheild delivered. A membrane will be inserted to the labial tunnel and tacked using 2 membrane tacks.
  Arms: Immediate implant placement with the bone shielding concept

SUMMARY:
Immediate implant placement has proven to be a successful treatment procedure that is preferred by patients because of being less traumatic, more time-efficient. Nowadays, the main goal of a successful immediate implant treatment has ceased to be gaining stability and osseointegration, but achieving long-term dimensional stability has become the optimal challenge. Various soft tissue and hard tissue augmentation techniques have been investigated in order to maintain the ridge dimensions following extraction and immediate implant placement.

DETAILED DESCRIPTION:
It has been noted that the different augmentation procedures aid in decreasing the dimensional changes occurring after immediate implant placement in the esthetic zone. Even though immediate implant placement is a predictable procedure, however, labial bone resorption following tooth extraction is inevitable. The available surgical techniques present do not entirely prevent dimensional variations of the peri-implant hard and soft tissues over time. Furthermore, substantial evidence showed that immediate implant placement failed to halt the resorption of the thin buccal bony plate with subsequent gingival recession, particularly in patients with thin gingival phenotype

ELIGIBILITY:
Inclusion Criteria:

* adult (>18 years) patients having a single non-adjacent hopeless maxillary tooth in the esthetic zone
* type I socket (intact but thin labial plate of bone and intact overlying soft tissues)
* adequate palatal bone
* ≥3 mm apical bone to engage the immediately placed implants
* optimum primary stability (a minimum of 30 Ncm insertion torque) following tooth extraction.

Exclusion Criteria:

* smokers
* pregnant women
* patients with systemic diseases
* periodontal disease, gingival recession
* infected sockets
* periapical pathosis and history of chemotherapy or radiotherapy within the past 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Pink Esthetic Score | 6 months
  Pink Esthetic Score 1-14 score PES

SECONDARY OUTCOMES:
labial bone thickness | 6 months
  radiographic CBCT
Peri-implant probing depth | 6 months
  mm
Implant failure | 6 months
  yes/No

CONTACTS AND LOCATIONS:
Overall Officials: Abdelsalam El Askary, Principal Investigator — private practice, Alexandria, Egypt; Noha A Ghallab, PhD, Study Chair — Professor in the department of oral Medicine & Periodontology, Cairo University; Nesma M shemais, PhD, Study Director — Lecturer in the department of oral Medicine & Periodontology, Cairo University
Locations (1):
- ElAskary dental center, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elaskary A, Ghallab N, Thabet A, Shemais N. The bone shielding versus dual-zone concept in treating thin-walled fresh extraction sockets with immediate implant placement: Soft and hard tissue changes. A randomized clinical trial. Clin Implant Dent Relat Res. 2024 Feb;26(1):66-77. doi: 10.1111/cid.13275. Epub 2023 Sep 5. PMID 37669913